CLINICAL TRIAL: NCT05425381
Title: Improving Social, Emotional, Behavioral, and Academic Functioning of Elementary School Students Through the Interconnected Systems Framework
Brief Title: Improving Social, Emotional, Behavioral, and Academic Functioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: East Carolina University (Other)
Collaborators: University of South Carolina (Other); Medical University of South Carolina (Other); University of Florida (Other)
Responsible Party: Principal Investigator, Brandon Kyle Schultz, Associate Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R324A210179
Record Dates: First submitted 2022-06-02; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Depression, Anxiety; Disruptive Behavior Disorder; Trauma, Psychological
Keywords: school mental health; interconnected systems framework
MeSH Terms: conditions — Depression; Anxiety Disorders; Attention Deficit and Disruptive Behavior Disorders; Psychological Trauma | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: The study will compare the ISFE model against co-located PBIS and SMH services-an approach commonly used in schools, particularly when community-based mental health clinicians are contracted for services. Thus, schools will be randomly assigned to the experimental conditions before systemic changes are implemented, beginning in the fall of 2022.
Who Masked: Participant
Masking Description: All student participants in the study will be assigned an alpha-numeric code to de-identify their cases. The codes and relevant identifiers will be maintained by a data specialist in the school districts and not shared with the researchers at any point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced version of Interconnected Systems Framework (ISFE) (Experimental): The ISFE addresses limitations of positive behavioral interventions and supports (PBIS) and school mental health (SMH) and improves the quality of services within the three tiers of multi-tiered systems of support (MTSS) by providing specific guidance on their systematic interconnection. Meaningful interconnection requires effective interdisciplinary collaboration, well-functioning teams, data-based decision making, and effective selection and implementation of evidence-based practices. The original interconnected systems framework (ISF) capitalizes on PBIS' strong implementation infrastructure and universal prevention strategies and combines these elements with SMH enhancements to Tiers 2 and 3 to achieve a comprehensive continuum of evidence-based practices. The ISFE leverages the strengths of PBIS and SMH to create one integrated system of care that achieves synergy and economies of scale.
  Interventions: Behavioral: Enhanced version of Interconnected Systems Framework
- Positive Behavioral Interventions and Supports with Co-located School Mental Health (PBIS+SMH) (Active Comparator): Mental health clinicians will be assigned and can work with MTSS teams (or not). Otherwise, there will be no special guidance. We expect this condition to mimic typical practices in schools, where PBIS and SMH efforts are co-located, but not meaningfully interconnected. In other words, we expect parallel functioning (Splett et al., 2014).
  Interventions: Behavioral: Positive Behavioral Interventions and Supports with Co-located School Mental Health

INTERVENTIONS:
Behavioral: Enhanced version of Interconnected Systems Framework — * District-community Leadership Team to support district-wide implementation and dissemination (Swain-Bradway et al., 2015)
  * Detailed memoranda of understanding between schools and collaborating mental health centers
  * Community mental health clinicians meaningfully participate in MTSS teams
  * Twice-monthly MTSS meetings using systematic teaming strategies (Newton et al., 2012)
  * Universal screening of students' social, emotional, behavioral, and academic functioning
  * Data-based decision-making using screening data and data on school and academic functioning for students with and without disabilities
  * Student-level discipline and intervention data (Blake et al., 2011; Smolkowski et al., 2016) addressed through iterative problem-solving approaches (McIntosh et al., 2018)
  * Team fidelity measures taken at the start and end of each school year, augmented with monthly fidelity monitoring of Tier 2 and 3 services
  * A Community of Practice (Wenger, 2010) among the ISFE schools
  Other Names: ISFE
  Arms: Enhanced version of Interconnected Systems Framework (ISFE)
Behavioral: Positive Behavioral Interventions and Supports with Co-located School Mental Health — * PBIS, including previously established data-based decision making, teaming, and evidence-based practices at three tiers: universal prevention; early identification and intervention for students with emerging risk; and intensive intervention for students with established problems and/or disabilities (Sugai & Horner, 2006; Sugai et al., 2014). Most PBIS schools struggle with intervention (Hawken et al., 2009) and the emphasis is typically on behavior, not internalizing student needs, including depression, anxiety, and trauma (Weist et al., 2018).
  * SMH using a co-located approach, with clinicians implementing treatment separate from the schools' MTSS (Barrett et al., 2013). Research has shown that even when PBIS and community-supported SMH operate in the same school building, in most cases there is no functional collaboration, (Splett et al., 2014). Under this model, SMH services are provided reactively, and students are often in crisis when referred (Dowdy et al., 2010).
  Other Names: PBIS+SMH
  Arms: Positive Behavioral Interventions and Supports with Co-located School Mental Health (PBIS+SMH)

SUMMARY:
This efficacy trial will evaluate the impact of an enhanced version of the Interconnected Systems Framework (ISFE) on elementary school-based team functioning, including use of evidence-based practices, and student emotional, behavioral, and academic functioning. The original interconnected systems framework (ISF) model was designed to improve the depth and quality of mental health services delivered within multi-tiered systems of support by integrating Positive Behavioral Interventions and Supports (PBIS) and school mental health (SMH) efforts to provide a continuum of high-quality services for students. Preliminary findings from a prior efficacy study show that the ISF improved team functioning and increased identification and services for students in need, particularly among youth of color, when compared to the other two conditions. Moreover, the ISF led to improvements in student social, emotional, and behavioral functioning. The current study builds on these findings by testing an enhanced version of the ISF designed to advance the model by adding/modifying several core components intended to further increase the impacts for youth with significant emotional and behavioral problems and reduce inequities in discipline and student service delivery.

DETAILED DESCRIPTION:
The Interconnected Systems Framework (ISF) for School Mental Health (SMH) and Positive Behavioral Interventions and Supports (PBIS) has been in development since 2009, involving leaders from national centers dedicated to both school mental health and positive behavioral support. The ISF was fully articulated in two widely disseminated monographs and is being implemented in more than 30 sites around the nation, supported by the national PBIS center (www.pbis.org), the Midwest PBIS network (www.midwestpbis.org), and other national networks focused on PBIS (e.g., www.midatlanticpbis.org, www.schoolbehavioralhealth.org). A recently completed randomized controlled trial (RCT) operating in 24 elementary schools (12 in Charleston, SC, and 12 in Marion, FL), funded by the National Institute of Justice (NIJ) tested the impact of the ISF as compared to PBIS alone, or PBIS with SMH clinicians, operating separately, which is the norm. In the current study, researchers will build from the previous findings to improve implementation efficacy and to better understand the change processes of the ISF. Specifically, researchers will test an ISF enhanced, or ISFE, based on lessons learned from the previous trial, and test its benefits for students with and without disabilities, while also exploring its impact in reducing inequities in discipline and service delivery for racial/ethnic minority youth.

Traditionally, ISF leverages the strengths of PBIS and school mental health to improve the quality of services across three tiers of prevention by providing specific guidance on their systematic interconnection. The ISF includes a district-community leadership team (DCLT), memoranda of agreement between schools and mental health providers, community-based clinicians integrated into problem-solving teams, universal social, emotional, and behavioral screening, team and intervention fidelity monitoring, and district-level communities of practice. The ISFE model tested in this study will have seven enhancements: (1) consistent meetings of the DCLT, which will include education, mental health, other youth-serving systems, and family/youth leaders; (2) clear agreements indicating parameters for an effective problem-solving team with community mental health clinician involvement; (3) improved team meeting procedures and data-based decision making with consistent use of a systematic program to facilitate comprehensive and efficient data review, decision-making, and follow through; (4) improved progress monitoring and fidelity monitoring of targeted and individualized interventions; (5) improved data-based decision making; (6) general enhancements to screening and measurement, including measures with strong psychometric properties; and (7) increased focus on, and better assessment of, student achievement, attendance, tardiness, grades, and discipline outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Elementary schools from pre-selected North Carolina (NC) and South Carolina (SC) school districts
* Serving K-5 students
* Comparable sociodemographic characteristics and fidelity of PBIS implementation
* Principals' consent to Participate
* Students from participating schools
* 3rd grade

Exclusion Criteria:

* Elementary schools from pre-selected NC and SC school districts
* Serving K-8 students
* Students from participating schools
* Children identified with a moderate or severe intellectual disability resulting in inability to participate in student self-report measures
* Children whose parents have submitted an opt-out form
* Children who opt out the day of data collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1208 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on Tiered Fidelity Inventory (TFI) for all Schools | Baseline; annually through study completion in first semester of each school year
  Tiered Fidelity Inventory (TFI) provides a valid, reliable, and efficient measure of the extent to which school personnel are applying the core features of school-wide positive behavioral interventions and supports.
Change Over Time on Interconnected Systems Framework Implementation Inventory (ISFII) for schools in the experimental condition | Once per semester in each intervention school year
  The ISFII was developed by the national Interconnected Systems Framework workgroup and includes 15 items for each of the three tiers. Early analyses support the tool's reliability, structural validity, and criterion-related validity as evidenced by strong correlations to similar measures at Tiers 2 and 3 (e.g., Benchmarks for Advanced Tiers; Anderson et al., 2009). The ISFII also appears to discriminate between schools showing some progress on ISF and those making few implementation efforts.
Change Over Time on Universal Fidelity Tool (UFT) for schools in the experimental condition | Monthly during intervention school years
  The UFT is a multi-dimensional, three-part measure for social, emotional, and behavioral interventions implemented in schools. The UFT measures intervention selection (the extent to which the intervention was selected based on data and matches identified problem areas), intervention delivery (the extent to which critical components of skill building, fluency, and maintenance are implemented during each session), and intervention monitoring (e.g., dosage, engagement, impacts). The UFT is a new measure with evidence for its reliability and social validity (Holmes et al., 2018).
Change Over Time on Team Functioning Measure for All Schools | Upon completion of specified meeting type within intervention school years, at least weekly
  For MTSS and child study team meetings in all schools the investigators will request documentation, with one professional designated per meeting to collect these data (e.g., school psychologist, counselor, MH clinician). A form for this purpose will document the meeting length (time), professionals attending and their disciplines (e.g., teacher, school psychologist, clinician, principal), family members/students attending, whether data were reviewed for intervention planning or refinement, and whether follow-up actions from the last meeting were discussed.
Change Over Time on Intervention Receipt Form (IRF) for All Schools | Monthly in intervention school years
  The IRF is a spreadsheet completed by all intervention providers (e.g., counselors, MH clinicians, teachers) documenting the referral problem, the intervention provided, and the frequency/dose of the intervention. An intervention identified on any IRF will be considered "quality" if it is an evidence-based practice that matches the referral problem. To determine if an intervention is evidence-based, the investigators will search relevant databases of evidence-based practices (e.g., What Works Clearinghouse).
Change from Baseline on BIMAS-2 Standard Form Teacher Ratings for All Schools | Baseline, once per semester in intervention school years, and once in follow-up year
  The Behavior Intervention Monitoring Assessment System-2 (BIMAS-2) is a nationally standardized and norm-referenced screening tool directly related to social, emotional, behavioral, and academic functioning in children and adolescents in grades pre-k to 12. Assessments are available for teachers, parents, clinicians, and self (age 12 and over). The BIMAS-2 Standard Form includes 34 items that comprise three problem behavior scales (conduct, negative, affect, and cognitive/attention) and two adaptive scales (social and academic functioning). Evidence of internal consistency, standard error of measurement, test-retest reliability, standard error of prediction, consistency between raters, and validity (content, convergent, divergent) is adequate to strong.
Change Over Time on BIMAS-2 Flex Assessment Teacher Ratings for All Schools | Baseline, once per semester in intervention school years, and once in follow-up year
  The Behavior Intervention Monitoring Assessment System-2 (BIMAS-2) is a nationally standardized and norm-referenced tool directly related to social, emotional, behavioral, and academic functioning in children and adolescents in grades pre-k to 12. Assessments are available for teachers, parents, clinicians, and self (age 12 and over). The BIMAS-2 provides change-sensitive Flex Assessments using a few (1-5) items that enable progress monitoring. This will be completed by teachers only for students referred to Tier 2 or Tier 3 assistance.
Change from Baseline on Student Self-Report Measures for All Schools | Baseline, once per semester in intervention school years, and once in follow-up year
  Combined version of the following rating scales: Brief Problem Checklist-12-item self-report for children 7-13 measuring internalizing and externalizing problems on a 3-point Likert scale Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Anxiety Subscale-8-item self-report measure for children 5-17 consisting of person-centered measures evaluating mental health PROMIS Pediatric Depression Subscale-8-item self-report measure for children 5-17 consisting of person-centered measures evaluating mental health PBIS School Climate Survey-11-item survey using a 4-point rating scale for grades 3-5 to assess students' perception of school climate along 4 dimensions: school connectedness, school safety, school orderliness, and peer and adult relations Social Emotional Health Survey-Primary- 20-item self-report measure using a 4-point Likert scale to assess adolescents' psychological strengths, including gratitude, zest, optimism, persistence, and prosocial behavior
Change Over Time in Student-level Achievement and School Records for All Schools | Once per school year through study completion
  Student reading and math achievement will be collected at both participating sites using i-Ready (Curriculum Associates, 2020), which the participating districts already administer three times each academic year. i-Ready identifies student strengths and weaknesses by assessing skills relative to grade-level expectations and standards, which allows progress monitoring at the student-level.
  Districts will provide academic records that include grades, absences, lateness, office discipline referrals, suspensions, and expulsions. The district will also report student entry into special education, increases/decreases in restrictiveness of special education programs, entry into alternative schools, and exit from special services.
Cost-Effectiveness of IFSE Condition Compared to PBIS+SMH Condition | Weekly during intervention school years
  An online tracking system will collect data relative to personnel, facilities, materials, equipment, and other inputs (e.g., special travel requirements). The tracking system will record personnel hours and activities, facilities usage, materials, equipment, and special travel, providing data for all major cost ingredients.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon K Schultz, Ed.D., Principal Investigator — East Carolina University; Mark D Weist, Ph.D., Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - East Carolina University, Greenville, North Carolina
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dowdy E, Ritchey K, Kamphaus RW. School-Based Screening: A Population-Based Approach to Inform and Monitor Children's Mental Health Needs. School Ment Health. 2010 Dec;2(4):166-176. doi: 10.1007/s12310-010-9036-3. Epub 2010 Apr 27. PMID 21088687
- [Background] Splett JW, Michael KD, Minard C, Stevens R, Johnson L, Reynolds H, Faerber K, Weist MD. State of the Carolinas: Implementing school mental health and Positive Behavioral Interventions and Supports. Rep Emot Behav Disord Youth, Special Issue. 2014; 14(4):87-95.
- [Background] Sugai G, Horner RR. A promising approach for expanding and sustaining school- wide positive behavior support. School Psych Rev. 2006;35(2):245.
- [Background] Sugai G, Simonsen B, Bradshaw C, Horner R, Lewis TJ. Delivering high quality school-wide positive behavior support in inclusive schools. In: McLeskey,J, Waldron, NL, Spooner, F, Algozzine, B, editors. Handbook of effective inclusive schools. New York: Routledge; 2014. P. 306-21.
- [Background] Hawken L, Adolphson S, Macleod K, Shuman J. Secondary-tier interventions and supports. In Sailor W, Dunlap G, Sugai G, Horner R, editors. Handbook of positive behavior support. New York: Springer; 2009. p. 395-420.
- [Background] Weist MD, Eber L, Horner R, Splett J, Putnam R, Barrett S, Perales K, Fairchild AJ, Hoover S. Improving multitiered systems of support for students with "internalizing" emotional/behavioral problems. J Posit Behav Interv. 2018 Jul; 20(3):172-84.
- [Background] Barrett S, Eber L, Weist MD. Advancing education effectiveness: An interconnected systems framework for Positive Behavioral Interventions and Supports (PBIS) and school mental health. Eugene (OR): University of Oregon Press; 2013. 189 p. Supported by the Center for Positive Behavioral Interventions and Supports (funded by the Office of Special Education Programs, US Department of Education).
- [Background] Anderson C, Childs K, Kincaid D, Horner RH, George H, Todd AW, Spaulding S. Benchmarks for advanced tiers. Eugene (OR): University of Oregon Educational and Community Supports; 2009.
- [Background] Holmes SR, Owens S, Reinke WM. Maximizing measurement: A universal and multidimensional approach to fidelity. Paper presented at: National Association of School Psychologists Annual Convention; 2018 Feb 13-16; Chicago, IL.
- [Background] McDougal JW, Bardos AN, Meier ST. Behavior Intervention Monitoring Assessment System: Technical manual. Toronto: Multi-Health Systems; 2011.